CLINICAL TRIAL: NCT06534307
Title: Langzeiteffekt Einer Pentaerithrityltetranitrat (PETN)-Behandlung in Der Schwangerschaft - Nachbeobachtung Der Kinder Der PETN-Studien
Brief Title: Long-term Follow-up of Children Born in the PETN Studies
Acronym: LOOP
Status: Recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Tanja Groten, Deputy Head of Department of Obstetrics, Jena University Hospital
Other Study IDs: ZKSJ0133
Record Dates: First submitted 2024-05-14; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Intrauterine Growth Restriction; Pentaerithrityl Teratnitrate in Pregnancy; Long-Term Effects to Children
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Physical Examination; Mass Screening; Electroencephalography; ABCB10 protein, human; 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Kidney Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — DNA-methylation and gene expression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Placebo: children of mothers that have been taken placebos during participation of PETN study
  Interventions: Behavioral: Questionnaire Child Behaviour Checklist; Behavioral: Questionnaire Young Self Report; Diagnostic Test: physical examination; Diagnostic Test: metabolic examination; Behavioral: Questionnaire Reynolds Intellectual Assessment Scales and Screening; Diagnostic Test: electroencephalogram; Other: Questionnaire Movement Assessment Battery for Children; Other: Questionnaire Continuous Performance Test; Other: Questionnaire Diagnostic System for Mental Disorders; Diagnostic Test: kidney function tests; Other: Questionnaire Five to Fifteen; Diagnostic Test: cardiovacular examination
- PETN: children of mothers that have been taken in PETN during participation of PETN study
  Interventions: Behavioral: Questionnaire Child Behaviour Checklist; Behavioral: Questionnaire Young Self Report; Diagnostic Test: physical examination; Diagnostic Test: metabolic examination; Behavioral: Questionnaire Reynolds Intellectual Assessment Scales and Screening; Diagnostic Test: electroencephalogram; Other: Questionnaire Movement Assessment Battery for Children; Other: Questionnaire Continuous Performance Test; Other: Questionnaire Diagnostic System for Mental Disorders; Diagnostic Test: kidney function tests; Other: Questionnaire Five to Fifteen; Diagnostic Test: cardiovacular examination

INTERVENTIONS:
Behavioral: Questionnaire Child Behaviour Checklist — The Child Behavior Checklist comprises items assigned to 8 subscales describing various behavioral areas. These subscales can be summed up to scores for internalizing and externalizing problems as well as a total score. Checklist scores are reported on a T-scale. Range of T-scale from scores 20 to 100 (average performance between scores 40 and 60). Higher scores mean higher amount of problems.
  Other Names: CBCL/6-18R
Behavioral: Questionnaire Young Self Report — The Questionnaire Young Self Report comprises items assigned to 8 subscales describing various behavioral areas. These subscales can be summed up to scores for internalizing and externalizing problems as well as a total score.
  Other Names: YSR/11-18R
Diagnostic Test: physical examination — physical development examination including height (in cm), weight (in g) and tanner states
Diagnostic Test: metabolic examination — metabolic development using blood analysis including blood components, metabolic parameters (Glucose, HbA1c, cholestrol)
Behavioral: Questionnaire Reynolds Intellectual Assessment Scales and Screening — The RIAS is standardized intelligence test. The RIAS provides an "Total Intelligence Index" (GIX, estimate of the general intelligence/g-factor), Verbal Intelligence Index (VIX) and the Nonverbal Intelligence Index (NIX). Test scores are reported on a T-scale. Range of T-scale from scores 20 to 100 (average performance between scores 40 and 60). Higher scores mean better cognitive performance.
  Other Names: RIAS
Diagnostic Test: electroencephalogram — neurocognitive development
  Other Names: EEG
Other: Questionnaire Movement Assessment Battery for Children — The M-ABC-2 is an standardized test to assess the motoric development. Adding up subscores addressing manual dexterity, aiming and catching, and balance delivers a total score of the motoric performance.
  Test scores are reported on a T-scale. Range of T-scale from scores 20 to 100 (average performance between scores 40 and 60). Higher scores mean better performance.
  Other Names: M-ABC-2
Other: Questionnaire Continuous Performance Test — The CPT measures selective attention, sustained attention as well as impulsive behavior. Checklist scores are reported on a T-scale. Range of T-scale from scores 20 to 100 (average performance between scores 40 and 60). Higher scores mean worse performance.
  Other Names: CPT
Other: Questionnaire Diagnostic System for Mental Disorders — The FBB-ADHS assesses a total score for ADHD-like behavior and subscores for the symptom trias of ADHD (attention deficit, motoric hyperactivity as well as impulsive behavior, Questionnaire scores are reported on a T-scale. Range of T-scale from scores 20 to 100 (average performance between scores 40 and 60). Higher scores mean higher amount of symptoms.
  Other Names: FBB-ADHS
Diagnostic Test: kidney function tests — urine examination (proteomics, cytokines, lipidomics)
Other: Questionnaire Five to Fifteen — The FTF 5-15R is a questionnaire to evaluate the child's developmental outcome in different areas of everyday life (cognition, language, and motor impairment as well as social, emotional, and behavioral problems). Individual item scores are added up per area and divided by the number of items. This results in a common scale value. Range of Percentile scores from 0 to 100 (0-90: no developmental problem; 90 and higher: hint for developmental problem). Higher scores mean worse developmental outcome.
  Other Names: FTF 5-15R
Diagnostic Test: cardiovacular examination — measurement of pulse wave velocity
  Other Names: Arteriograph

SUMMARY:
In every 10th pregnancy, the child in the uterus is insufficiently nourished, a so-called growth retardation. This occurs when the child cannot reach its growth potential due to an undersupply in the uterus. This inadequate supply is considered a developmental cause for the later development of physical diseases like cardiovascular diseases, sugar metabolism disorders and obesity as well as mental developmental problems (for example problems in cognitive skills, deficits in language development, concentration and attention).

From 2002 to 2008, 111 patients with impaired placental blood flow were included in a small study and treated with Pentalong or placebo. From 2017 to 2022, the positive effects of the study treatment were tested on a larger number of patients. A total of 317 pregnant women were included at 14 participating study centers in Germany.

In this follow-up study, the development of the children born in the two studies will be examined. The study consists of two independent parts: firstly, questionnaires are answered by the former participants and secondly, an on-site visit is carried out to check the physical and mental health of the child.

DETAILED DESCRIPTION:
Pregnancies in which impaired uterine blood flow is detected by Doppler measurements during routine examinations in the second trimester are at high risk of developing fetal growth restriction (FGR). FGR affects 10% of pregnancies and is the leading cause of perinatal mortality and morbidity. In addition, intrauterine growth restriction places a lifelong burden on the physical and mental health of affected children. Epidemiological studies have shown that children with FGR have an increased risk of developing type 2 diabetes mellitus, hypertension, dyslipidemia and a high BMI. In addition, the affected children show disorders in hormonal balance and pubertal development as well as specific impairments of various cognitive and neurocognitive functions. There is also a link between FGR and lower cognitive ability in preschool children, school-age children and young adults, as well as lower communication, language and reading skills in school-age children. Neuronal development (e.g. EEG frequency spectra, resting-state networks) and executive functions are also impaired by FGR.

In the follow-up study, the children will be examined from the age of 6. Here, the effects of PETN on the development of children of women with high-risk pregnancies can be further investigated and a comparative study of growth-retarded and normal-growth children can also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* mothers participation in one of the PETN studies
* age above 5 years
* completion of questionnaires for self reported data
* written consent for physical examination

Exclusion Criteria - only physical examination:

* physical and mental states preventing physical examination

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all live born children from participants of the PETN-studies
Sampling Method: Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
childrens behaviour | up to 2 years after study inclusion
  total score of either CBCL/16-18R or YSR/11-18R

SECONDARY OUTCOMES:
physical development height | up to 2 years after study inclusion
  height of the child in cm
physical development weight | up to 2 years after study inclusion
  weight of the child in kg
age appropriate development | up to 2 years after study inclusion
  age appropriate development documented as "yes or no" question in german routine examination plan ("Kinderuntersuchungsheft") in the last 6 years at caregivers
cognitive, motoric, and exectuve function | up to 2 years after study inclusion
  scores of the eight domains of the FTF 5-15-R
physical development | age above 10 years
  self reported tanner states
cardiovascular development | age of 6 to 8 years
  pulse wave velosity
IQ development | age of 6 to 8 years
  scores of RIAS test
motoric development | age of 6 to 8 years
  total score of M-ABC-2
attention behaviour | age of 6 to 8 years
  scores of the four domains of the cpt
symptoms of attention and activity disorders | age of 6 to 8 years
  total scores of DISYPS-III
neurocognitive development | age of 6 to 8 years
  results of EEG power measurement in alpha band
neurocognitive development | age of 6 to 8 years
  results of EEG power measurement in beta band
neurocognitive development | age of 6 to 8 years
  results of EEG power measurement in gamma band
neurocognitive development | age of 6 to 8 years
  results of EEG power measurement in delta band
neurocognitive development | age of 6 to 8 years
  results of EEG power measurement in theta band
epigenetic analysis | age of 6 to 8 years
  DNA-methylation

CONTACTS AND LOCATIONS:
Locations (13):
- Germany (13):
  - Universitäts-Frauenklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Städtisches Klinikum München, München, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Uniklinikum Leipzig, Leipzig, Saxony
  - Krankenhaus St. Elisabeth und St. Barbara, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Berlin Charité Campus Mitte, Berlin
  - Berlin Vivantes Klinikum Neukölln, Berlin

IPD SHARING:
Plan to Share IPD: No